CLINICAL TRIAL: NCT02730533
Title: The Efficacy of Esomeprazole Premedication on Intraoperative Bleeding During Gastric ESD: an Endoscopist-blinded Randomized Controlled Study
Brief Title: The Efficacy of Esomeprazole Premedication on Intraoperative Bleeding During Gastric ESD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Zhiguo Liu, Associate Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY20162024-1
Record Dates: First submitted 2016-03-28; First posted 2016-04-06 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Stomach Neoplasms
Keywords: endoscopic submucosal dissection; proton pump inhibitor; bleeding
MeSH Terms: conditions — Stomach Neoplasms; Hemorrhage | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (Active Comparator): No PPI treatment should given after the initial allocation. Patient will be admitted, and ESD will be performed. Then a 3-day i.v. treatment of esomeprazole will be initiated after ESD procedure and followed by a 26 days oral treatment with esomeprazole tablets 40 mg.
  Interventions: Drug: No PPI treatment
- Esomeprazole group (Experimental): Esomeprazole should start as soon as possible after the initial allocation. During the 7 days of p.o. treatment, patient will be admitted, and ESD will be performed as soon as completing the p.o. treatment. Then a 3-day i.v. treatment of esomeprazole will be initiated after ESD procedure and followed by a 26 days oral treatment with esomeprazole tablets 40 mg.
  Interventions: Drug: Esomeprazole

INTERVENTIONS:
Drug: Esomeprazole — Proton pump inhibitor
  Arms: Esomeprazole group
Drug: No PPI treatment — No PPI treatment before ESD procedure
  Arms: Control group

SUMMARY:
This will be a single-centre, randomised, endoscopist-blind, parallel-group study in patients who are scheduled endoscopic submucosal dissection (ESD) for gastric mucosal lesion. The primary objective is to observe whether a regimen of 7-day oral esomeprazole premedication can alleviate intraoperative bleeding in patients scheduled for ESD due to gastric mucosal lesions.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and the willingness to sign a written informed consent document.
* Female or male aged ≥18 years.
* Patients must have gastric mucosal lesion that are eligible for ESD indications (Japanese Gastric Cancer Association 2011), including early gastric cancer, polyps, adenoma, and precancerous/suspected lesions diagnosed by endoscopy.

Exclusion Criteria:

* Malignancy or other advanced disease with a life expectancy of < 6 months as judged by the investigator.
* The ASA classification of physical status ≥ 4 as judged by the investigator.
* Severe hepatic disease or renal disease
* Ability to understand and the willingness to sign a written informed consent document.
* Major cardiovascular event at enrollment or within 3 months prior to enrollment such as stroke, myocardial infarction, or hospitalization for treatment of unstable angina pectoris as judged by the investigator.
* Haemorrhagic disorder.
* Patients who had a history of gastrectomy or a recurrent lesion.
* Known or suspected hypersensitivity to any component of any PPI .
* Planned treatment with: warfarin (including other vitamin K antagonists), cisapride, phenytoin, atazanavir, nelfinavir, digoxin, methotrexate, clopidogrel, tacrolimus, theophylline, lidocaine, nifedipine.
* Pregnancy, planned pregnancy or lactation. Women of childbearing potential must use reliable and medically accepted methods of birth control, as judged by the investigator.
* Known or suspected alcohol, drug or medication abuse.
* Any condition associated with poor compliance as judged by the investigator.
* Participation in any study involving administration of an investigational product or device within the preceding 14 days prior to enrollment.
* Involvement in the planning and conduct of the study. Previous enrollment in the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The total bleeding rate according to grading of intraoperative bleeding during ESD procedure | 1 day
  ≥grade 1 means bleeding

SECONDARY OUTCOMES:
The frequency of coagrasper usage which reflects grade of major bleeding | 1 day
Post-ESD ulcer quality as indicated in description | 1 day
  Ulcer base quality will be evaluated base on the grading of clean, with minor trace of coagulation, base with extensive coagulation.
Intra-procedure injury to muscularis propria including perforation. | 1 day
  Injury of muscularis propria will be evaluated as no injury, minor injury and deep injury/perforation.
Mean haemoglobin reduction between intervention and control group. | 1 day
Delayed bleeding rate as indicated by haematemesis and melaena | 30 days
The mean percentage of mucosal defect reduction at follow-up endoscopy on 28 days after ESD procedure. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Zhiguo Liu, Principal Investigator — Xijing Hospital of Digestive Disease
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Paper publishing

REFERENCES:
- [Background] Ahn JY, Jung HY, Choi KD, Choi JY, Kim MY, Lee JH, Choi KS, Kim DH, Song HJ, Lee GH, Kim JH, Park YS. Endoscopic and oncologic outcomes after endoscopic resection for early gastric cancer: 1370 cases of absolute and extended indications. Gastrointest Endosc. 2011 Sep;74(3):485-93. doi: 10.1016/j.gie.2011.04.038. Epub 2011 Jul 13. PMID 21741645
- [Background] Choi MK, Kim GH, Park DY, Song GA, Kim DU, Ryu DY, Lee BE, Cheong JH, Cho M. Long-term outcomes of endoscopic submucosal dissection for early gastric cancer: a single-center experience. Surg Endosc. 2013 Nov;27(11):4250-8. doi: 10.1007/s00464-013-3030-4. Epub 2013 Jun 14. PMID 23765426
- [Background] Deprez PH, Bergman JJ, Meisner S, Ponchon T, Repici A, Dinis-Ribeiro M, Haringsma J. Current practice with endoscopic submucosal dissection in Europe: position statement from a panel of experts. Endoscopy. 2010 Oct;42(10):853-8. doi: 10.1055/s-0030-1255563. Epub 2010 Jul 9. PMID 20623442
- [Background] Fujishiro M, Chiu PW, Wang HP. Role of antisecretory agents for gastric endoscopic submucosal dissection. Dig Endosc. 2013 Mar;25 Suppl 1:86-93. doi: 10.1111/j.1443-1661.2012.01370.x. Epub 2013 Jan 24. PMID 23368844
- [Background] Gotoda T, Kondo H, Ono H, Saito Y, Yamaguchi H, Saito D, Yokota T. A new endoscopic mucosal resection procedure using an insulation-tipped electrosurgical knife for rectal flat lesions: report of two cases. Gastrointest Endosc. 1999 Oct;50(4):560-3. doi: 10.1016/s0016-5107(99)70084-2. No abstract available. PMID 10502182
- [Background] Jang JS, Choi SR, Graham DY, Kwon HC, Kim MC, Jeong JS, Won JJ, Han SY, Noh MH, Lee JH, Lee SW, Baek YH, Kim MJ, Jeong DS, Kim SK. Risk factors for immediate and delayed bleeding associated with endoscopic submucosal dissection of gastric neoplastic lesions. Scand J Gastroenterol. 2009;44(11):1370-6. doi: 10.3109/00365520903194609. PMID 19891589